CLINICAL TRIAL: NCT02164383
Title: A Quit Smoking Study Using Smartphones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-1606; P50CA143188 (NIH)
Record Dates: First submitted 2014-06-11; First posted 2014-06-16 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-03

CONDITIONS: Smoking Cessation; Smoking; Nicotine Dependence
Keywords: Smoking Cessation; Smoking; Nicotine
MeSH Terms: conditions — Smoking Cessation; Smoking; Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mobile Games (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? Nicotine patch plus behavioral cessation counseling with access to Mobile Games.
  Interventions: Drug: Nicotine patch; Behavioral: Cessation Counseling; Device: Mobile Games
- No Mobile Games (Experimental): This arm of the project will address the following question:
  How effective is the following intervention:
  Nicotine patch plus behavioral cessation counseling without access to Mobile Games.
  Interventions: Drug: Nicotine patch; Behavioral: Cessation Counseling

INTERVENTIONS:
Drug: Nicotine patch — 4-week starter kit of nicotine patch
Behavioral: Cessation Counseling — 5 brief counseling sessions
Device: Mobile Games
  Arms: Mobile Games

SUMMARY:
The objective of this research is to determine whether smartphone games show promise for helping smokers increase their chances of quitting. The central hypothesis is that smokers who have access to smartphone games during their quit smoking attempt will smoke fewer cigarettes and report less craving than will smokers without such access.

ELIGIBILITY:
Inclusion Criteria:

* being age 18 or older;
* being able to read and write English;
* being willing and able to learn how to use a smartphone if they have not used one before;
* smoking 10 or more cigarettes per day for the past 6 months;
* having an expired carbon monoxide rating of 6 ppm or greater;
* not having been diagnosed with or treated for schizophrenia, psychosis or bipolar disorder in the past 10 years;
* being willing to make a quit attempt in 2 weeks;
* agreeing to attend clinic visits, receive coaching calls, and complete brief smartphone assessments;
* planning to remain in the area for at least the next 2 months;
* using the following alternative tobacco products (a pipe, full sized cigars, snuff or chew) no more than two times a week over the past month;
* being willing to stop using electronic cigarettes (e-cigarettes) for the 6 weeks they are in the study;
* not currently taking bupropion, Wellbutrin, or Zyban;
* if currently using nicotine replacement therapy or Varenicline, agreeing to use only study medication for the duration of the study;
* being willing and able to use the nicotine patch;
* never having had a serious skin reaction or other allergic reaction to the nicotine patch;
* not pregnant, trying to conceive, or nursing;
* if a woman of childbearing potential, agreeing to use or having their partner use an acceptable method of birth control during a 2 month period (1 month of nicotine patch and 1 month after). (Acceptable methods of birth control include: abstinence, condoms, diaphragm, birth control pills or injectable contraceptive [e.g., Depo-Provera], an intrauterine device, hysterectomy, tubal ligation, sterilization, vasectomy, or being more than 2 years post-menopausal.)
* Participants need to report playing video games for no more than 60 minutes a day.
* Although participants can play console games, they need to be willing to not play any mobile games for 6 weeks during the study if they are asked to do so.
* Participants need to report being willing to stay in the study even if they are not at first successful in quitting smoking.
* They need to report that they have a way to get to the clinic.

Exclusion Criteria:

* They will be excluded if in the last 4 weeks they have been hospitalized for any of the following: a stroke, heart attack, congestive heart failure, or an abnormal electrocardiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya R. Schlam, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Schlam TR, Baker TB. Playing Around with Quitting Smoking: A Randomized Pilot Trial of Mobile Games as a Craving Response Strategy. Games Health J. 2020 Feb;9(1):64-70. doi: 10.1089/g4h.2019.0030. Epub 2019 Sep 19. PMID 31536384

RESULTS

PARTICIPANT FLOW:
Groups:
- Mobile Games: This arm of the project will address the following question:
  How effective is the following intervention? Nicotine patch plus behavioral cessation counseling with access to Mobile Games.
  Nicotine patch: 4-week starter kit of nicotine patch
  Cessation Counseling: 5 brief counseling sessions
  Mobile Games
- No Mobile Games: This arm of the project will address the following question:
  How effective is the following intervention:
  Nicotine patch plus behavioral cessation counseling without access to Mobile Games.
  Nicotine patch: 4-week starter kit of nicotine patch
  Cessation Counseling: 5 brief counseling sessions
Period: Overall Study
Arm/Group | Mobile Games | No Mobile Games
Started | 16 | 14
Completed | 15 | 14
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Games | No Mobile Games | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.06 (10.27) | 43.79 (13.50) | 40.73 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 14 | 29
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 14 | 13 | 27
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change Between Baseline Mean Cigarettes Smoked Per Day and Mean Cigarettes Smoked Per Day During the First 4 Weeks of the Quit Attempt Calculated as Percentage Change
Description: Every day participants will report the number of cigarettes they smoked that day at baseline and for the first 4 weeks of the quit attempt (starting on the target quit day) using timeline followback assessment. This information will be used to calculate a participant's change in mean cigarettes smoked per day from baseline compared to the mean across the first 4 weeks of the quit attempt calculated as percentage change.
Time Frame: Cigarettes per day measured daily for the first 4 weeks of the quit attempt (starting on the target quit day) and at baseline
Measure: Mean (Standard Deviation); unit: percentage change in cigarettes per day
Arm/Group | Mobile Games | No Mobile Games
Number analyzed (Participants) | 16 | 14
percentage change in cigarettes per day | -86.08 (22.06) | -84.26 (30.03)
Statistical Analysis 1: Comparison: Mobile Games vs No Mobile Games; Test type: Superiority; p = .85, ANOVA; Mean Difference (Final Values) = 1.82 — ANOVA results: F(1,28)=.04, p=.85, partial eta-squared (as a measure of effect size) = .001

ADVERSE EVENTS:
Time Frame: Adverse event data were collected 3 times during one month of treatment.
Description: Participants were asked "Since your last contact with us, have there been any changes in your medical condition or health?" on the target quit day (TQD), 2 weeks post-TQD, and 4 weeks post-TQD. Only nicotine-related adverse events were counted. A total of 15 nicotine-related adverse events were assessed.
Arm/Group | Mobile Games | No Mobile Games
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 1/16 | 2/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mobile Games (N=16) | No Mobile Games (N=14)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Itching or hives (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No